CLINICAL TRIAL: NCT03596710
Title: Radiologically Guided Biopsies of Metastatic Castration Resistant Prostate Cancer to Identify Adaptive Mechanisms of Resistance in Patients Undergoing 177Lu-PSMA Radioligand Therapy
Brief Title: Image-Guided Biopsies in Identifying Mechanisms of Resistance in Participants With Metastatic Castration Resistant Prostate Cancer Undergoing Radioligand Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor withdrew study
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-000273; NCI-2018-01422 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18-000273 (Other: UCLA / Jonsson Comprehensive Cancer Center); P50CA092131 (NIH)
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2018-07

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Image-Guided Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (image-guided biopsy) (Experimental): Participants undergo image-guided biopsy over 45 minutes prior to first RLT course and 1-2 days after the third RLT course.
  Interventions: Procedure: Image Guided Biopsy

INTERVENTIONS:
Procedure: Image Guided Biopsy — Undergo image guided biopsy
  Other Names: Image-Guided Biopsy; Imaging Guided Biopsy

SUMMARY:
This trial studies image-guided biopsies work in identifying mechanisms of resistance in participants with castration resistant prostate cancer that has spread to other places in the body and who are undergoing radioligand therapy (RLT). Tissue sample collected from a biopsy may help determine why response to RLT varies among patients, and this may help researchers to find better treatments for advanced prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Proportion of metastatic castration resistant prostate cancer (mCRPC) patients with altered signaling pathways after radioligand therapy assessed by phospho-proteomics of biopsy samples.

SECONDARY OBJECTIVES:

I. Generation of patient derived xenograft (PDX) models to determine if tumor levels of activity for individual adaptive pathways are related to the best prostate specific antigen (PSA) response.

II. Sequencing to identify frequently mutated genes such as TP53 and ATM.

OUTLINE:

Participants undergo image-guided biopsy over 45 minutes prior to first RLT course and 1-2 days after the third RLT course.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer patient
* Histologically confirmed prostate cancer
* Enrolled in Lu-PSMA-617 treatment trial (Institutional Review Board [IRB]# 17-000330)
* Based on positron emission tomography (PET)/computed tomography (CT) images: evidence of lymph node or soft tissue metastatic disease amenable to image-guided biopsy
* Platelets > 75,000/ul within 14 days prior to biopsy
* Prothrombin time (PT) or international normalized ratio (INR) and a partial thromboplastin time (PTT) < 1.5 times the institutional upper limit of normal (ULN) within 14 days prior to biopsy
* Patients on warfarin, aspirin, or other anti-coagulants are eligible provided they are deemed able to tolerate discontinuation of anti-coagulation for one week prior to the biopsy. Conversion to low molecular weight heparin prior to biopsy is permitted per local standard operating procedures, provided there is agreement regarding the procedure between the treating physician, the interventional radiologist and the principal investigator (PI)

Exclusion Criteria:

* Patients with significant congenital or acquired bleeding disorders (e.g. von Wildebrand's disease, acquired bleeding factor inhibitors) are not eligible

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2021-06-14 (Estimated); Study Completion 2022-06-14 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a successful evaluable biopsy with altered signaling pathways after radioligand therapy (RLT) | Up to 3 years
  No statistical power analysis was performed as this is a pilot study. An unbiased proteomic/phospho-proteomics analysis will be done and it is unknown how many and which parameters will change in response to radioligand therapy. The study will in subsequent studies use the information obtained here to design a more definitive trial.

SECONDARY OUTCOMES:
Proportion of patients with gene mutation in regulators of replication stress response according to sequencing | Up to 3 years
  No statistical power analysis was performed as this is a pilot study. An unbiased proteomic/phospho-proteomics analysis will be done and it is unknown how many and which parameters will change in response to radioligand therapy. The study will in subsequent studies use the information obtained here to design a more definitive trial.
Generation of xenografts | Up to 3 years
  No statistical power analysis was performed as this is a pilot study. An unbiased proteomic/phospho-proteomics analysis will be done and it is unknown how many and which parameters will change in response to radioligand therapy. The study will in subsequent studies use the information obtained here to design a more definitive trial.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Rettig, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center